CLINICAL TRIAL: NCT06987422
Title: Investigation of Plantar Fascia and Achilles Tendon Thickness and Flexibility in Individuals With Pes Planus
Brief Title: Plantar Fascia and Achilles Tendon Thickness and Flexibility in Pes Planus
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Busra Seckinogullari Korkusuz, Principal Investigator, Ankara University
Other Study IDs: 604.01.02-421
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-07

CONDITIONS: Pes Planus
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pes Planus: Individuals with pes planus
- Control: Healthy individuals with similar demographic characteristics

SUMMARY:
The aim of this study is to examine the plantar fascia and Achilles tendon thickness and flexibility in individuals with pes planus. Individuals between the ages of 18-45 who have been diagnosed with pes planus by an orthopedist and healthy individuals with similar demographic characteristics will be included in the study as a control group. Demographic information of the individuals will be recorded and clinical evaluations will be made. The foot posture of the individuals participating in the study will be evaluated with the Foot Posture Index, and the degree of flat feet will be evaluated with the Navicular Drop Test. The Achilles tendon and plantar fascia thicknesses of the individuals participating in the study will be measured with ultrasound, and the plantar fascia and Achilles tendon flexibility will be measured with a myotonometer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45
* Mini Mental State Examination (MMSE) score of 24 to 30
* Diagnosed with Pes Planus by a physician

Exclusion Criteria:

* Inability to communicate verbally
* Use of walking aids
* Any history of surgery involving the lower extremities
* People with severe visual impairment, neurological disorders and/or congestive heart failure.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals with Pes Planus
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2025-05-25 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Foot Posture Index | Baseline
  In this study, the Foot Posture Index will be used to evaluate the foot postures of the participants.
Navicular Drop Test | Baseline
  The Navicular Drop Test will be administered to measure the amount of drop in the participants' navicular bones.
Ultrasonographic Evaluation | Baseline
  Participants' Achilles tendon and plantar fascia thicknesses will be evaluated using a high-resolution ultrasound device.
Myotonometer | Baseline
  Participants' plantar fascia and Achilles tendon flexibility will be evaluated using a myotonometer device.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Korkusuz, PhD, Study Chair — Atılım University; Büşra Seçkinoğulları Korkusuz, PhD, Principal Investigator — Ankara University
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Angin S, Crofts G, Mickle KJ, Nester CJ. Ultrasound evaluation of foot muscles and plantar fascia in pes planus. Gait Posture. 2014;40(1):48-52. doi: 10.1016/j.gaitpost.2014.02.008. Epub 2014 Feb 26. PMID 24630465
- [Result] Tas S, Aktas A, Dikici TF, Cekok FK. Achilles Tendon, Patellar Tendon, and Femoral Cartilage Thickness in Control vs Asymptomatic Flatfoot Young Adults. Foot Ankle Int. 2023 Jan;44(1):81-88. doi: 10.1177/10711007221136137. Epub 2022 Nov 22. PMID 36412188